CLINICAL TRIAL: NCT07269899
Title: A Phase I Study Evaluating the Preliminary Efficacy and Safety of WTX212A Injection as Monotherapy or in Combination With Radiotherapy in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of WTX212A Monotherapy or in Combination With Radiotherapy in Patients With Advanced Solid Tumors
Acronym: Reboot-107
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Westlake Therapeutics (Industry)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, Principal Investigator, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Reboot-107
Record Dates: First submitted 2025-08-12; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor Cancer; Cancer
Keywords: Solid Tumor Cancer; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Number of Cohort : 2
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Cohort A (Experimental): Experimental: Cohort A Intervention: Drug: WTX212A Monotherapy
  Interventions: Drug: WTX212A injection
- Experimental: Cohort B (Experimental): Experimental: Cohort B Intervention: Drug: WTX212A+Radiotherapy
  Interventions: Drug: WTX212A injection; Radiation: radiotherapy

INTERVENTIONS:
Drug: WTX212A injection — Erythrocyte-αPD-1 Antibody Conjugates
  Other Names: Erythrocyte-αPD-1 Antibody Conjugates
Radiation: radiotherapy — Radiotherapy will be administered sequentially, with WTX212A treatment starting within one week after the completion of radiotherapy
  Arms: Experimental: Cohort B

SUMMARY:
This is a single-arm, open-label, investigator-initiated clinical study (IIT) designed to evaluate the preliminary efficacy, safety, tolerability, immunogenicity, and pharmacokinetic (PK) characteristics of WTX212A Injection in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a single-arm, open-label, investigator-initiated clinical study (IIT) designed to evaluate the preliminary efficacy, safety, tolerability, immunogenicity, and pharmacokinetic (PK) characteristics of WTX212A Injection in patients with advanced solid tumors. The study is divided into two phases: an initial exploratory phase and an expansion phase. The study includes two cohorts: Cohort A (WTX212A monotherapy) and Cohort B (WTX212A in combination with radiotherapy)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent, understanding of the study, and willingness and ability to complete all study procedures.
2. Male or female, aged 18 to 75 years (inclusive).
3. Patients with histologically and/or cytologically confirmed advanced malignant tumors.

Exclusion Criteria:

1. Suffering from other serious internal diseases, including but not limited to: uncontrolled diabetes, active peptic ulcer, liver cirrhosis, active bleeding, etc., those with uncontrollable or severe cardiovascular diseases, such as NYHA Class II or higher congestive heart failure, unstable angina, myocardial infarction, etc., within 6 months before the first dose, difficult to control hypertension (systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥100mmHg).
2. Uncontrollable pleural effusion, peritoneal effusion, or pericardial effusion requiring puncture and drainage, or recurrence requiring re-drainage after puncture and drainage.
3. History of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, or severe lung function impairment.
4. Previous IO drug treatment with adverse events related to the drug that required permanent discontinuation of IO treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of WTX212A monotherapy or WTX212A in combination with radiotherapy | From enrollment to the end of treatment，an average of 1 year
  Objective Response Rate (ORR) of WTX212A monotherapy or WTX212A in combination with radiotherapy
Efficacy of WTX212A monotherapy or WTX212A in combination with radiotherapy | From enrollment to the end of treatment，an average of 1 year
  Disease Control Rate (DCR) of WTX212A monotherapy or WTX212A in combination with radiotherapy

SECONDARY OUTCOMES:
Efficacy of WTX212A monotherapy or WTX212A in combination with radiotherapy | Every 6 weeks until the end of the last treatment ，an average of 1 year
  Progression-Free Survival (PFS).etc of WTX212A monotherapy or WTX212A in combination with radiotherapy, as evaluated using the Evaluation Criteria in Solid Tumors (Version 1.1).
Safety of WTX212A monotherapy or WTX212A in combination with radiotherapy | From the first treatment to the end of the safety visit，an average of 1 year
  Incidence of adverse events (AEs), treatment-related AEs, and serious adverse events (SAEs) of WTX212A monotherapy or WTX212A in combination with radiotherapy.
Pharmacokinetic characteristics(Cmax) | Through study completion, an average of 1 year
  Pharmacokinetic parameters of peripheral blood in subjects after administration, including but not limited to Cmax
Pharmacokinetic characteristics(Tmax) | Through study completion, an average of 1 year
  Pharmacokinetic parameters of peripheral blood in subjects after administration, including but not limited to Tmax
Pharmacokinetic characteristics(AUC0-t) | Through study completion, an average of 1 year
  Pharmacokinetic parameters of peripheral blood in subjects after administration, including but not limited to AUC0-t
Pharmacokinetic characteristics(t1/2) | Through study completion, an average of 1 year
  Pharmacokinetic parameters of peripheral blood in subjects after administration, including but not limited to t1/2
Pharmacokinetic characteristics(CL) | Through study completion, an average of 1 year
  Pharmacokinetic parameters of peripheral blood in subjects after administration, including but not limited to CL
Number of Anti-drug antibody (ADA) | Through study completion, an average of 1 year
  Describe the number of anti-drug antibodies (ADA) produced by subjects at each time point after treatment, and the time of producing ADA.
Percentage of Anti-drug antibody (ADA) | Through study completion, an average of 1 year
  Describe the percentage of anti-drug antibodies (ADA) produced by subjects at each time point after treatment, and the time of producing ADA.

OTHER OUTCOMES:
Assess Biomarkers Relevant to the Study（T-Cell) | Through study completion, an average of 1 year
  Assess the percentages of immune cell subsets (T-Cell ) before and after treatment for advanced malignant tumors, changes in immunophenotyping and other meaningful Biomarkers
Assess Biomarkers Relevant to the Study（MDSC) | Through study completion, an average of 1 year
  Assess the percentages of MDSC before and after treatment for advanced malignant tumors, changes in immunophenotyping and other meaningful Biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: RuiHua Xu, PhD, Principal Investigator — Cancer Center of SUN YAT-senU
Locations (2):
- China (2):
  - Cancer Center of SUN YAT-senU, Guangzhou, Guangdong
  - Cancer center of Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided